CLINICAL TRIAL: NCT06412731
Title: Comparing the Effectiveness of Papain Based Chemico-mechanical Caries Removal Gel and 38% Silver Diamine Fluoride for Treating Active Caries Lesion of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Alhamzah thaer hasan Ankaz, BDS, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUPRU004
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries in Children
Keywords: CMCR; SDF; Ceramic bur
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ceramic bur (Cerabur) C (Active Comparator): Cera bur (Ceramic Bur) Komet, Lemgo, Germany
  Interventions: Other: Cera-bur
- Silver Diamine Fluoride (e-SDF) S (Active Comparator): e-SDF (SDF 38%) E-kids, India
  Interventions: Other: E-SDF
- CMCR gel (Brix3000) B (Active Comparator): Brix3000 (Papain based gel) S.R.L., Argentina
  Interventions: Other: Brix3000

INTERVENTIONS:
Other: Cera-bur — Dental caries removal using a low-speed handpiece and a ceramic bur and restoring the cavity with Glass ionomer filling material
  Other Names: Ceramic bur
  Arms: Ceramic bur (Cerabur) C
Other: Brix3000 — Chemical-dissolving active dental caries and hand instrument used for removing the lesion then restoring with Glass ionomer filling material
  Other Names: Papain-based CMCR
  Arms: CMCR gel (Brix3000) B
Other: E-SDF — Arresting the infected dentin and the demineralized lesion covered with Glass-ionomer filling
  Other Names: 38% Silver Diamine fluoride
  Arms: Silver Diamine Fluoride (e-SDF) S

SUMMARY:
This study aims to investigate the efficacy of silver diamine fluoride (SDF) and Papain-based chemico-mechanical caries removal gel and using ceramic bur as a control in treating dentine caries in primary molars aged 7-8 years children. by investigating the following outcomes:

1. Arrestment of caries lesion and the emergence of a new one
2. Time required for the treatment
3. Adverse events
4. Children's anxiety

DETAILED DESCRIPTION:
The traditional approach to removing caries with dental burs is the most often used technique in the treatment of dental caries. However, this method is continuously associated with many disadvantages, such as patients finding drilling uncomfortable, the frequent need for local anesthetic, and detrimental heat effects on the pulp.

The purpose of this research was to evaluate three minimally invasive therapies via the assessment of:

1. Duration of treatment
2. (feeling of pain) and the need for anesthetic
3. Incidents with negative outcomes that have been officially documented
4. Filling material adhesiveness fellow up

The null hypothesis was that there was no difference among Silver Diamine Fluoride, Brix3000 Papain based Chemico-mechanical caries removal product, and ceramic burr in time, anxiety, and pain, reported side effect

Randomized control clinical trial will be allocated into 3 groups: S group (treatment with SDF), B group (treatment with Brix3000 Papain based gel), and C group as control (treatment by rotary handpiece Smart bur)

Setting:

Sample collection: the samples are to be collected at The College of Dentistry, Al-Mustansiriyah University - Iraq- Baghdad Subject The sample size will be 45 children aged 7-8 years with primary molars with occlusal active caries lesions.

ELIGIBILITY:
Inclusion Criteria:

* Each child should have primary molars with open carious lesions, either on the occlusal surface or Proximal one with the absence of a neighboring tooth.
* These lesions should affect the dentin but not expose the pulp.
* The depth of the cavities should measure between 40-99 using a DIAGNOdent caries detection instrument for standardization

Exclusion Criteria:

* Children were excluded if parents were unwilling to be assigned to any of the approaches
* Children that had any abnormal medical condition or silver or papain allergy
* Chose molars with clinical or radiographic signals of pulp involvement

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Adverse event | during the first two weeks
  The following adverse events will be investigated: Pain, sensitivity, tooth discoloration, burning in the mouth, allergy altered taste of food, irritation of the gums or mucosa
Filling fellow up | after 3 months
  The evaluation was done using the community periodontal index (CPI)-probe (WHO-probe) and a dental mirror. The treated lesions were classified according to the evaluation scores which were modified from those used by Francis et al.: score 1 - the restoration intact, covering all pits and fissures; score 2 - the restoration partially lost, the tooth is sound (no active/soft caries); score 3 - the restoration partially lost, the tooth is carious(active/soft caries); score 4 - the restoration completely lost, the tooth is sound; and score 5 - the restoration completely lost, the tooth is carious. The tooth was considered sound if its surface felt hard and shiny

SECONDARY OUTCOMES:
anxiety level | immediately after the procedure
  Anxiety level prescribed by the patient using a facial image scale to measure the children' anxiety. Each kid was instructed to indicate the facial expression that most accurately conveyed their current emotional state, which may be categorized as either (very happy; happy; neutral; unhappy; or very unhappy
Time | This will take about from 5 to 30 minutes
  the time required for the treatment in each group using a digital timer A digital timer which triggers as soon as the tooth brushing starts. During the first appointment starting from dental caries removal until sound dentin reached before Glass ionomer filling placement,

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Mustansiriyah University, Baghdad, Al-karkh, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satyarup D, Mohanty S, Nagarajappa R, Mahapatra I, Dalai RP. Comparison of the effectiveness of 38% silver diamine fluoride and atraumatic restorative treatment for treating dental caries in a school setting: A randomized clinical trial. Dent Med Probl. 2022 Apr-Jun;59(2):217-223. doi: 10.17219/dmp/143547. PMID 35506381
- [Background] Vollu AL, Rodrigues GF, Rougemount Teixeira RV, Cruz LR, Dos Santos Massa G, de Lima Moreira JP, Luiz RR, Barja-Fidalgo F, Fonseca-Goncalves A. Efficacy of 30% silver diamine fluoride compared to atraumatic restorative treatment on dentine caries arrestment in primary molars of preschool children: A 12-months parallel randomized controlled clinical trial. J Dent. 2019 Sep;88:103165. doi: 10.1016/j.jdent.2019.07.003. Epub 2019 Jul 4. PMID 31279925
- See also: Comparative Evaluation of 'Less Invasive Approach' of caries excavation and 'Only Arrest And No Excavation Approach' in dental caries management in primary molars- A Randomised Controlled Trial — https://jamdsr.com/uploadfiles/17vol9issue8pp84-92.20210815050049.pdf
- See also: Evaluation of the Efficacy of Caries Removal Using Papain Gel (Brix 3000) and Smart Preparation Bur(in vivo Comparative Study) — https://global-ie.com/wp-content/uploads/2022/02/comparativo-brix-vs-fresas-inteligentes.pdf